CLINICAL TRIAL: NCT06405360
Title: DEUX OEUFs:Cracking the Potential of Eggs to Improve Child Growth and Development
Brief Title: DEUX OEUFs: Cracking the Potential of Eggs to Improve Child Growth and Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: World Vision (Other); University of Rwanda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UFlorida 202301484
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Infant Malnutrition; Fetal Growth Retardation
Keywords: Nutrition; Maternal Health; Infant growth and development; Maternal diet
MeSH Terms: conditions — Infant Nutrition Disorders; Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcomes assessors will be blinded to the intervention arm once the participant is enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Mothers in the intervention arm will receive an animal-source food supplement of two eggs per day from the day of enrollment during the first trimester through childbirth.
  Interventions: Dietary Supplement: Egg consumption
- Control Arm (No Intervention): Mothers in the control arm will be asked to continue consuming their typical diet

INTERVENTIONS:
Dietary Supplement: Egg consumption — Participants in the intervention group will be provided two eggs to consume daily.
  Arms: Intervention Arm

SUMMARY:
This proposed randomized controlled trial aims to investigate the effect of maternal egg consumption during pregnancy on birth length. The study hypothesizes that mothers who consume two eggs a day will have children whose birth length is significantly longer than those born to mothers who consume a typical diet. Pregnant women (n=956) from Nyagatare District in Rwanda will be randomized into one of two study arms: a treatment group (T1) or a control group (T2). Mothers in the treatment arm will receive an animal source food (ASF) supplement of two eggs per day, from enrollment during first trimester through childbirth. Mothers in the control arm will be asked to continue consuming their typical diet. Mothers in both arms will receive standard information, education, and communication about health and nutrition during pregnancy and after birth. All enrolled mothers in the study will also receive up- to-date standard care for pregnant women, as outlined by the Government of Rwanda, a fortified blended flour if they are not already receiving it from the government, a mobile phone with cellular connection, health insurance if they do not already have, and compensation for traveling to a Community Health Worker's home every day for study engagement. All women will receive ultrasound examinations three times during pregnancy, as well as blood tests for anemia. Women in the control arm will receive additional compensation at childbirth. Women will be recruited and enrolled during first trimester (9-14 weeks gestational age), as confirmed by ultrasound. At enrollment, baseline data will be collected on socio-economic factors, maternal health, maternal diet, and fetal growth. Additional markers for maternal health and child growth and development, including markers for fetal brain development, will be collected during two targeted ante-natal clinic visits (20-26 weeks and 30-34 weeks), where all women will receive ultrasound assessment in addition to their typical clinical assessment. At childbirth, maternal and child health data will be collected, including birth outcomes, child anthropometry, and indicators of neurodevelopment. Additional follow-up of maternal and child health indicators, including maternal depression, and infant and young child feeding practices, will be collected at 1 month and 6 months of child age.

DETAILED DESCRIPTION:
Background and Significance

Inadequate and less diverse diets during critical life stages including pregnancy, lactation, and infancy contribute to malnutrition of children, particularly in low- and middle-income countries (LMICs) The first thousand days post-conception has been identified as a critical period of potential intervention within which to reduce stunting and improve early childhood development. Maternal nutritional status has been shown to directly affect the occurrence of child stunting, as well as indirectly affect stunting through other child factors. The use of WHO child growth standards has revealed that intrauterine growth faltering is a greater problem than previously realized and that pediatric growth faltering often begins in utero and is directly related to maternal nutrition.

Maternal diets have an important role to play in overall maternal and child health, as maternal nutrition is an important predictor of pregnancy outcomes, fetal growth and development, and birth outcomes. The increase in nutritional demands during pregnancy and lactation is well established.

In LMICs, typical diets are less diverse and often lack animal source foods (ASF), which are a rich source of bioavailable macro and micronutrients. The nutritional value of ASF has been highlighted as an important dietary tool in efforts to reduce child malnutrition due to high nutrient density and bioavailability of macronutrients, as well as essential micronutrients, which may be suboptimal in vegetarian diets. Given these nutritional advantages when compared to plant based diets, there is an increasing dialogue around efforts to increase ASF in the diet, low rate particularly in smallholder farming communities in LMICs, where dietary diversity is typically low and nutritional outcomes are poor. However, a recent Cochrane review found insufficient evidence to indicate that ASF was more effective than plant-based diets in improving child growth, pointing explicitly to the need for trials that are adequately powered and that study specific ASF.

Eggs are an excellent source of protein, essential fatty acids, and vitamins A and B12, as well as choline and docosahexaenoic acid (DHA), nutrients associated with child growth and cognitive development. Like other ASF across LMIC, eggs are rarely consumed among populations of women of reproductive age in sub-Saharan African, particularly in rural areas where rates of malnutrition are high, despite the relative affordability and availability of eggs compared to other ASF. Recent research indicates that upon the introduction of complementary foods, the consumption of eggs by infants and young children may improve nutritional outcomes in LMICs.

To date, studies that examined eggs as a dietary tool with which to reduce malnutrition have focused on child egg consumption (at 6 months of age or later), with little to no research exploring the potential impact of nutritional interventions that target consumption of eggs among pregnant or lactating mothers as a mechanism to improve both maternal and child health outcomes. Given the alignment of nutrient demand during pregnancy and the nutrient composition and bioavailability in ASF, this study hypothesizes that consumption of ASF during pregnancy will improve fetal growth in areas where malnutrition is prevalent. To the study's knowledge, no study has focused solely on maternal ASF consumption during pregnancy to investigate its impact on fetal growth and child health outcomes. This randomized control trial will address an existing gap in the literature surrounding the potential effect of maternal consumption of a specific ASF (eggs) on in-utero growth faltering and brain development.

Hypotheses, Aims, and Objectives/research questions :

H01: No significant difference will be observed between the length of children born to mothers who consume two eggs per day and those children born to mothers who consume a typical diet.

H11: Mothers who consume two eggs a day will have children whose birth length is significantly longer than those born to mothers who consume a typical diet Primary aim: The study will test the effects of a maternal nutritional intervention of two eggs per day, comparing child birth length of infants born to those women with infants born to women who consume a typical diet in Nyagatare District, Rwanda.

Methods Study Description:

This study is a randomized controlled trial that will examine the nutritional benefits of maternal egg consumption from the first trimester of pregnancy through childbirth, on child growth and development in Nyagatare District, Rwanda. Specifically, the study is powered to detect the difference in child birth length between those born to mothers who received two eggs a day throughout pregnancy and those consuming the typical diet for the district. Women will receive the nutritional supplement through childbirth. They will be monitored during four clinic visits within this time period (enrollment at first trimester, second trimester, third trimester, and childbirth). The mother and infant will then stay enrolled in the study for follow up at one month and six months postpartum. In addition to birth length (primary outcome), the study will also investigate effects of the nutritional intervention on in-utero brain development, newborn developmental assessment, six month LAZ, and six month developmental assessment. 956 pregnant women will be recruited and independently assigned to one of the two research arms.

Study Design:

All enrolled mothers will be randomized into one of two study arms: a treatment group (T1) or a control group (T2). Mothers in the treatment arm will receive an ASF supplement of two eggs per day, from the day of enrollment during first trimester through childbirth. Mothers in the control arm will be asked to continue consuming their typical diet. Mothers in both arms will receive standard information, education, and communication about healthy diet during pregnancy, and will not be restricted from adding eggs or any other food to their diet. Mothers in both arms will

receive standard information, education, and communication about healthy diet during pregnancy, and will not be restricted from adding eggs or any other food to their diet. All enrolled mothers in the study will receive the up-to-date GoR standard care for pregnant women, a mobile phone with cellular connection, health insurance (if not already covered), and compensation for traveling to a CHW's home every day for study engagement. Any enrolled mother not receiving 6 kg of Shisha Kibondo (SK) per month, per GoR standard of care for mothers who are undernourished, will receive during pregnancy 6 kg/month of a fortified flour (CSB+) that is nutritionally comparable to SK. Dietary supplements will be initiated upon enrollment and will continue through childbirth; target enrollment is first trimester (9-<14 weeks' gestation). Participants will include mother-child dyads: pregnant women will be recruited, enrolled, and followed, with their children, for the first six months of the child's life. Health risks attributed to egg consumption have historically been associated with the high cholesterol content in eggs and possible increased risk of cardiovascular disease (CVD). However, results are inconclusive in the existing literature, and almost all published research is on populations in high income countries. Consequently, it has been suggested that, where evident, the harmful effects of eggs may be attributed to negative dietary patterns associated with high levels of food intake rather than egg consumption. While there is mixed evidence on the overall health benefits and risk of egg consumption in the general population, increasingly, science supports consumption of eggs as part of a healthy diet. Prior to intervention, study staff will inquire with participants about any known reaction or allergies to eggs. Past reaction or allergy to egg consumption will render the participant ineligible to participate. The study will carefully document and report any adverse reactions to egg consumption.

Study Site and Study Population: The intervention will take place in Nyagatare District in Eastern Province, Rwanda, and specifically the catchment areas of Ndama and Karangazi Health Centers. Please note, if enrollment pace does not align with expectations, which are based on formative research and published numbers of births, then expanding enrollment and intervention preparation to a third health center will be considered.

Intervention :

This study will have one intervention arm and one control arm - provision of two eggs daily during pregnancy, or typical diet. Eggs will be prepared daily at Karangazi and/or Ndama Health Centers by trained study personnel and according to quality control procedures that ensure daily preparation and serving is safe (described below). Eggs will be fully cooked (boiled or steamed) and prepared with clean water. The study team will provide cooking pots, cooking fuel, and stoves, as well as cleaning supplies and clean water with which to wash pots, and additional storage and serving utensils as needed at food preparation centers.

Following preparation, a Food Distributor will be used to coordinate transporting eggs daily to village-based distribution points, which will be CHW homes. The study will transport eggs from preparation centers to the villages of enrolled mothers. Motos will be equipped with shelving support to transport eggs such that they remain intact and safe for consumption. CSB+ packages will be distributed to all the women. Procurement will be done directly from the manufacturer of Shisha Kibondo, to ensure comparability of that which is received by mothers enrolled in the GoR program and by the study.

All women enrolled in the study will be asked to visit a designated village- based consumption site (CHW home) daily. Women in the treatment arm will receive eggs and nutrition and health messaging at the site at a designated time of day, women in the control arm will receive only nutritional messaging and will be asked to come during a different window of time. Sites will be located within an approximately 20-minute walk from women's homes; if no site is available within this radius, additional distribution sites will be identified as needed. Women in each intervention arm will be asked to come during separate times or meet in separate locations to minimize spillover between the treatment and control arms. All women (intervention and control) will be compensated for their daily travel to the CHW's house. Current plans are to compensate women at 500 RWF per day IF they come at least 6 days in a week. This amount or threshold may change slightly following piloting, based on community acceptability. In order to increase acceptability and adherence of egg consumption, salt will be available to accompany egg consumption. Women will receive eggs by CHWs and their consumption will be directly observed and recorded (including whether partial or complete consumption) by CHWs, local volunteers trained by WV, or study staff. Confirmation of the woman's identification will be ensured through use of photos (taken during active consumption), daily sign-in, and use of a study participant ID card and/or phone scan.

CHWs will receive a prorated monthly compensation of 30,000 RWF for their participation and support in the study. In situations where the CHWs are unavailable due to other duties or travel, a WV volunteer will distribute eggs and observe egg consumption. In situations where CHW absence is unavoidable, the study staff will work closely with the CHW and will use the CHW's home, if possible, for distribution. Only when that is not possible an alternative distribution site will be identified for those particular days and women will be kept abreast of these changes by use of study provided cell phones. Adherence to the intervention will be monitored throughout the study to ensure high uptake, with the goal of 100% adherence (daily observed consumption of 2 eggs per day, 7 days a week). Although 100% adherence is desired, the study team recognizes that the woman may not present on certain days due to travel outside of the study area, work or family obligations, sickness, or other reasons. The woman also has the option of refusing the food on any given day. If and when a mother fails to present to the study team to receive her assigned supplement without a prior notification of absence or explanation, a team member will attempt to contact the mother and visit again later in the day in an effort to ensure adherence. At the end of the day, however, if a mother has not come to the CHW home to receive the eggs, WV staff may travel to her home to try to deliver and observe egg consumption. This will occur any day that the woman does not present at the CHW home for egg consumption during the designated window. If nausea is identified as a barrier to daily consumption of the nutrition supplement, an over-the-counter (commercially available) anti- nausea medication will be provided. (Note: no antinausea medication provided will include any antihistamine). If the woman is hospitalized and remains within the study catchment area, the study team will deliver to the facility, with permission of health facility staff. Additionally, if the mother has not taken the food supplement due to absence, refusal, or other reason, but has not formally withdrawn from the study, the study team will attempt to contact the mother by phone or staff CHW outreach every 2-4 days to inquire about resuming the intervention for a period of 1 month. If the mother re-engages with the study team, all intervention and data collection will be reinstated. Any barriers to participation identified during the study will be considered and addressed, as possible, by the research team. If there is a loss of pregnancy, the woman will continue to receive the intervention for a period of 30 days.

Food safety: The project will ensure that the following conditions are met during the cycle of egg and CSB+ procurement and distribution; during egg preparation; and that all actors in food distribution are trained on the following aspects: QC processes (SOPs, monitoring, record keeping, etc.) for the distribution of eggs will be certified by the certification body in Rwanda which is Rwanda Standards Board (RSB). During the storage of eggs and CSB

+ from suppliers, the designated food handler will ensure that the storage location fulfills the required standards. Eggs will be stored for a maximum of 3 weeks. The CSB+ will be stored in a cool dry place and expiration dates will be monitored per manufacturer's guidelines. Lot numbers will be monitored and stored in case of product recall. Container for storage will be clean and dry.

Hygiene practices are observed and ensured during the provision of eggs to mothers.

Selection of Study Population Randomization procedure:

The study will individually randomize on a 1:1 basis, using stratified block randomization with varying block sizes to randomly assign the treatment arms to preserve the balance of treatments across enrollment locations (Ndama and Karangazi) and gestational age groups (9-11 weeks and 12-<14 weeks). The participants will be first stratified based on enrollment location and gestational age. A chain of blocks will be pre-generated for each stratum, e.g., 1000 blocks.

The size of each block will be randomly and independently chosen as 2, 4 or 6 individuals. Within each block of a given size, there are equal numbers of either arms but the order is randomly shuffled. For example, the first four blocks for a given site and a given gestational age group may look like [EGG (E), CONTROL (C), C, E]-[ CL, E]-[E, C]-[ CL, E, E CL, CL, E]. The first 14 patients will get the sequential assignments as in the chain. The team will use the tool at sealedenvelope.com to generate the randomization list. The random seed will be generated using the random integer generator at random.org which introduces randomness from unpredictable atmospheric noise. Each study site will receive its own randomization list. Each assignment will be stored in a sealed envelope, and envelopes will be ordered according to the randomization list in each gestational age group. When a study subject is screened for enrollment and is deemed eligible, she will be offered enrollment and engaged in an informed consent process. If she agrees to participate (consents), she will choose an envelope that has a piece of paper that indicates whether she is in the treatment (egg) or control (typical diet) group. Each individual subject will have a unique randomization code, in addition to a unique study ID, so that the original assignment of each subject can be easily tracked. Data analysts who will perform the actual analysis will be blinded about treatment assignments. The envelopes will be pre-filled in advance, and both the study participant and the staff person facilitating this randomization reveal process will be blinded to what is inside the envelope, until it is opened.

Study Procedures :

Before the enrollment begins, study staff will organize educational campaigns in the villages to promote early antenatal care visits (ANC ) visits and facilitate visits to health centers. Urine pregnancy tests will be distributed to CHWs to encourage confirmation of suspected pregnancy and attendance at a first antenatal care visit as early as possible to identify pregnancies as early as possible. At the commencement of the study, staff will coordinate with CHWs to compensate transportation costs for women with positive pregnancy tests from the village to the health care center serving the catchment area. On designated recruitment days, study staff will be available at the healthcare center to conduct standardized screening ultrasound and gather baseline data, as described below.

All pregnant women aged 18 years to 44 years (reported or based on ID card if available) with no plans to move outside the study area will be considered for enrollment as per eligibility criteria above. Study staff will perform an initial eligibility screening (including a urine pregnancy test if they haven't already had confirmation), administer informed consent, and conduct an ultrasound screening and eligibility confirmation. All ultrasounds will be conducted by OBGYNs engaged in the project or trained Nurse Sonographers. The pregnancy will be dated during the ultrasound screening using a validated AI-based algorithm (SCANNAV FetalCheck, IntelligentUltrasound, UK). Crown rump length (CRL) and head circumference will also be measured, in conjunction with reported last menstrual period (LMP) based on standard methods and INTERGROWTH 21st standards. Any fetal anomalies, extrauterine pregnancies, missed abortions, or other incidental abnormal findings will be referred to local healthcare facilities for appropriate care. CRL and head circumference-based dataing will be compared to AI-based gestational age dating based on ultrasound analysis. Women with confirmed pregnancy between 9 and <14 weeks will be invited to voluntarily participate in the study with appropriate informed written consent. Women who are below 9 weeks will be asked to return at a later date in order to meet eligibility criteria. Written consent will be read out loud to women as needed for low literacy. Based on current birth and delivery rates in the catchment area, enrollment of eligible pregnant women will start in May 2024 and is estimated to be complete by September 2025.

At the time of the enrollment, a baseline survey will be conducted on demographic and baseline characteristics of the household, livestock ownership, WASH, (socio-demographics), pregnancy and medical history, maternal behavior towards risk factors (Malaria), depression (psychosocial health), physical activity, dietary diversity, gender-based violence and household food security (See Baseline Questionnaire). Phone contact information on the study participant, other household members, and another acquaintance will be collected in order to ensure the study team can reach the study participant and child after birth. The study will measure the pregnant woman's height, weight, and mid upper arm circumference (MUAC). Standing height will be measured in duplicate using a stadiometer, with weight measured to nearest 0.1 kg using a digital scale (e.g., Seca). Resting blood pressure will be measured in triplicate, using a validated system (e.g., Omron) with appropriate cuff size based on the mother's MUAC.

After completion of the survey and anthropometric measures, the woman will be asked to provide a hair sample and will have a blood sample drawn by a trained phlebotomist. Maternal hemoglobin will be measured using a bioanalyzer to obtain a complete blood count analysis. The blood will be kept in a cooler box with ice packs and after isolating the serum will be put into a -20C cooler within 8 hours of collection. Within 7 days of collection, the sample will be transferred to Kigali for longer term storage in -80C freezers at the National Reference Lab (NRL) or similar facility.

Following the baseline survey, collection of anthropometric data, and blood sample, mothers will have a photo taken and will be registered as study participants. They will have a digital ID card created specific to the study, with barcode and photo, using WV's Last Mile Mobile Solutions (LMMS) platform. Following registration, women will be randomly allocated to the control arm or the two-egg daily arm, by selection of an envelope of their choice.

Following randomization, the chosen arm assignment will be added to the digital ID. A hard copy of the study participation card will be printed and laminated. The participant will be informed they need to present their study ID card at all health facility visits (including ANC visits and delivery, as well district/provincial hospital if there are complications). Furthermore, women in control and intervention will be instructed to sign-in and present their card each day at the designated distribution point in the village in order to receive the appropriate control or intervention content. Women who have a positive pregnancy test and are believed to be in their first trimester and are consented for eligibility screening will be given a 3000 RWF cash for participation regardless of final eligibility. If the mother is enrolled into the study and not currently enrolled in a health insurance scheme, study staff will facilitate and cover costs for enrollment for the mother and her family. CHWs will be compensated 30000 RWF monthly (prorated) for their efforts and involvement in enrollment, referrals, intervention delivery, and follow-up activities of the study.

Procedures for Second and Third Trimester Assessments (ANC Visits)

Participants will be asked to return to the health center monthly for their normal ANC visit schedules. At two of these ANC visits, the participant will be asked to engage following the ANC visit in additional study visits: one at 20-26 weeks and another at 30-34 weeks. They will also receive a text/phone call reminder of the study visit before each visit. At these visits, an OBGYN or nurse sonographer will conduct ultrasound measurements to assess fetal growth using fundal height and ultrasound imaging for brain development. Using the ultrasound machine, the trained sonographer will collect standard images for prenatal care, including: biparietal diameter; head circumference; cerebellar diameter; abdominal circumference; femur length; humerus length; and estimated fetal weight. The following additional measures will be taken: thalamic measurements in multiple dimensions and projections; corpus callosum length; and gangliothalamic ovoid measurements, including diameter, sagittal length and estimated volume. Images collected in the field will be shared with the research team for ongoing supervision and data quality monitoring. Fetal anomalies or other adverse conditions identified through ultrasound scanning will be referred to the appropriate medical facilities for care. At the 20-26 week and 30-34 week visit, participants will be asked to provide a hair sample, and maternal blood will be drawn and maternal hemoglobin measured as described above. Information on medical conditions since last visit, physical activity, breastfeeding intention and maternal diet will be collected using a short survey (See Pregnancy visit questionnaire). Anthropometric measurements will also be collected during the two ANC visits. All participants will receive 3000 RWF cash for attending these visits to compensate for their time.

Procedures for Birth Visit

All birth outcomes data will be collected up to 72 hours after birth, with the first 24 hours as the target window. Participants will notify study staff when they travel to a health facility for delivery, or if they are delivering at home. Study staff will also maintain communication with CHWs to stay updated regarding labor and delivery status. Birth outcomes will be measured by a trained study nurse. In the case of a home birth that doesn't report to the health center (expected to be approximately ><5-10% of deliveries), the Nurse Enumerator team will visit the house and conduct measurements there, with attention to ensuring as flat and safe a measurement environment as possible. Primary outcome birth length will be measured at the time of birth (<72hrs).

Two study Nurse Enumerators will together measure length in triplicate using length boards (Seca), to nearest 0.1 cm. Birth Weight will be measured to the nearest 0.1kg, using a digital scale (Seca). Head circumference of the infant will be measured to the nearest 0.1cm. Clinical characteristics of the birth and all antenatal care and postnatal visits (through 6 months of age) will be based on medical records (where consented) as well as maternal recall, including HIV status, who attended the birth, birth injury, and Apgar score. Blood will be drawn from the newborn at birth and stored as described above. At birth all enrolled women will receive an umbrella and to compensate for time for birth measures, 3000 RWF for a facility-based visit, and 1000 RWF for a home-based visit, depending on where the measures are conducted. Control women will additionally receive kitenge cloth at birth.

Procedures for Maternal and Child Follow-up Visits (1MO AND 6MO post-birth) After birth, there will be two follow-up visits at approximately 1 month and 6 months of age. All mother-child dyads will be visited by the study enumerators at their residence. At each of these visits, the mother or primary caregiver will answer a survey on each visit to document their own personal diet (DQQ), infant feeding practices, and whether the infant is exclusively breastfed (WHO IYCF, DQQ). The questionnaire will use WHO-recommended core indicators of optimal breast-feeding that includes early initiation of breastfeeding (within 1 h of birth), exclusive breastfeeding (EBF) till 6 months after birth. A survey module on the infant's health and morbidity (diarrhea, respiratory, fever, malaria) and care-seeking behavior will also be administered. If consented and pending funding availability, medical records at health facilities (outpatient, IMCI, inpatient) and CHW sick child encounter forms will be extracted to understand impacts of the nutrition interventions on child health outcomes, including diarrhea, respiratory infections, fever, and malaria, as well as mortality. The study will also administer survey questions regarding exposure to gender-based violence (using questions from the DHS), given associations with adverse birth outcomes and nutrition. Child length will be measured in triplicate using length boards (Seca), to nearest 0.1 cm. Weight will be measured to the nearest 0.1kg, using a digital scale (Seca). Head circumference of the infant will be measured to the nearest 0.1cm. MUAC will also be assessed, and referrals will be made for those classified as moderate or severe acute malnutrition. Additionally at 6 months of age, infants will be assessed for neurodevelopment using CREDI, a validated assessment tool that has been used previously in Rwanda. The CREDI (long-form) provides domain-specific scores in motor, cognitive, language, social-emotional development, as well as an overall score. Blood will be drawn from the infant at birth, and from both mother and infant at 1 month and 6 months, and stored as described below. Hair sample from mother will be requested, if consented. All participants will receive 1000 RWF cash for attending these visits to compensate for their time.

Sample size:

Studies with nutritional intervention during pregnancy have found a mean difference in LAZ ranging from 0.12, 0.19 to 0.29. However, there is no study that specifically looks at the impact of eggs or other ASF supplementation alone during pregnancy. Based on the available literature on other food supplementation and as found in some literature review papers, the study hypothesizes a mean difference of 0.18 in LAZ to be a reasonable and clinically meaningful effect size of a food-based intervention on birth length compared to a control arm. The sample size required with 20% attrition (accounting for pregnancy loss, stillbirths, and loss of follow-up) to attain an 80% marginal power with 5% level of significance was 478 per arm. Thus, the study aims to enroll an overall sample of 956 women in the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Lives in study area (catchment area of Karangazi Health Center and Ndama Health Center)
* Confirmed viable intrauterine pregnancy (confirmed via ultrasound)
* Aged between 18-44 years
* 9-14 weeks gestation (confirmed via ultrasound, up to 13 weeks +6 days)
* Agrees to participate with informed consent

Exclusion Criteria:

* Intention to move outside the study area in next 12 months
* Intention to deliver at a location outside of Eastern Province Nyagatare District
* Any known adverse reaction to eating eggs or porridge ingredients
* Any condition that could affect the ability to comply with the study requirements or understand the informed consent process
* Participation in other clinical trials (to avoid burden and potential interactions between interventions)
* Any individual unable or unwilling to comply with the study requirements, such as attending regular follow-up visits or adhering to prescribed nutritional supplementation.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 464 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Newborn Length for age z-score | Within 72 hours of birth
  Child's recumbent length at birth, standardized using the INTERGROWTH 21st growth standard

SECONDARY OUTCOMES:
Head circumference Z-scores | Between 20-26 weeks and 30-34 weeks gestational ages
  Ultrasound derived estimate of head circumference in cm (standardized using the INTERGROWTH 21st growth standards)
Femur length Z-scores | Between 20-26 weeks and 30-34 weeks gestational ages
  Ultrasound derived measure of femur length in cm (standardized using the INTERGROWTH 21st growth standards)
Abdominal circumference Z-scores | Between 20-26 weeks and 30-34 weeks gestational ages
  Ultrasound derived measure of abdominal circumference in cm (standardized using the INTERGROWTH 21st growth standards)
Biparietal Z-scores | Between 20-26 weeks and 30-34 weeks gestational ages
  Ultrasound derived biparietal diameter in cm (standardized using the INTERGROWTH 21st growth standards)
Estimated fetal weight Z-scores | Between 20-26 weeks and 30-34 weeks gestational ages
  Ultrasound derived fetal weight in g (standardized using the INTERGROWTH 21st growth standards)
Cerebellar diameter | Between 20-26 weeks and 30-34 weeks gestational ages
  Cerebellar diameter (axial plane) in cm, based on ultrasound
Corpus callosum length | Between 20-26 weeks and 30-34 weeks gestational ages
  Corpus callosum length in cm, based on ultrasound
Thalamus midline axial | Between 20-26 weeks and 30-34 weeks gestational ages
  Thalamic measurements in cm, based on ultrasound
Gangliothalamic ovoid diameter | Between 20-26 weeks and 30-34 weeks gestational ages
  Gangliothalamic ovoid diameter in cm, based on ultrasound
Gangliothalamic ovoid sagittal length | Between 20-26 weeks and 30-34 weeks gestational ages
  Gangliothalamic ovoid sagittal length in cm, based on ultrasound
Gangliothalamic ovoid estimated volume | Between 20-26 weeks and 30-34 weeks gestational ages
  Gangliothalamic ovoid estimated volume cubic cm, based on ultrasound
Gestational duration | At birth of newborn
  Gestational age in weeks at birth (among live births)
Preterm birth | At birth of newborn
  Proportion of live births <37 weeks completed gestation
Birthweight | Within 72 hours of birth
  Birthweight (g) among live births
Low birthweight | Within 72 hours of birth
  Proportion of live births that are low birthweight (<2500 g)
Birthweight for gestational age | Within 72 hours of birth
  Birth weight-for-age z-score according to INTERGROWTH 21st growth standards
Small for Gestational Age (SGA) at birth | Within 72 hours of birth
  Birthweight for gestational age at birth (10th percentile and 3rd percentile), according to INTERGROWTH 21st growth standards)
Small vulnerable newborn status among live births | Within 72 hours of birth
  Defined as SGA (10th percentile) according to INTERGROWTH 21st growth standards, preterm birth (<37 weeks completed gestation), or low birth weight <2500g
Newborn developmental assessment | At one month of age
  Hammersmith Neonatal Neurological Examination (HNNE)
Head circumference of newborn | Within 72 hours of birth
  Head circumference and head circumference z-score according to INTERGROWTH 21st growth standard
Maternal weight | Weight will be collected at enrolment (between 9-<14 weeks gestation), 20-26 weeks gestation, 30-34 weeks gestation, and during labor/delivery
  Maternal weight in kg
Maternal weight gain during pregnancy | Weight will be collected at enrolment (between 9-<14 weeks gestation), 20-26 weeks gestation, 30-34 weeks gestation, and during labor/delivery
  Designation of inadequate, adequate, and excessive weight gain according to IOM guidelines and calculated based on maternal weight at labor/delivery visit - maternal weight at enrolment.
Maternal cortisol concentration | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, at time of birth, and at 1 and 6 months post birth
  Cortisol concentration from maternal hair and/or nail samples (per participant preference)
Minimum Dietary Diversity for Women | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, and at 1 and 6 months post birth
  Dietary Quality Questionnaire will be used to generate the MDD-W, used here as meeting the validated threshold or not 0-10 scale, higher is more diversity (better) with threshold of having at least 5 to have met minimum requirements (coded as 0 for not having met/1 for have met MDD)
Dietary Diversity Score | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, and at 1 and 6 months post birth
  Dietary Quality Questionnaire will be used to generate the MDD-W, used here to generate a score (0-10), where 10 is highest dietary diversity
Maternal Hemoglobin | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, at time of birth, and at 1 and 6 months post birth
  We will measure hemoglobin, as indicated by trimester specific WHO cutoffs.
Maternal depression | At 6 weeks and 6 months post birth
  Edinburgh Postnatal Depression Scale (range 0-30; 12 or higher defining maternal depression)
Infant Length-for-age z-score | At 6 weeks and 6 months of age
  Length-for-age z-score according to the WHO Multicentre Growth Reference Study standard
Prevalence of Stunting among infants | At 6 weeks and 6 months of age
  Length-for-age z-score <-2 SD of the median according to the WHO Multicentre Growth Reference Study standard
Infant weight-for-age Z score | At 6 weeks and 6 months of age
  Weight-for-age Z score according to WHO standard
Prevalence of Underweight among infants | At 6 weeks and 6 months of age
  Weight-for-age z-score <-2 SD of the median according to the WHO Multicentre Growth Reference Study standard
Child neurodevelopment | 6 months of age
  Measured according to the Caregiver Reported Early Childhood Development Instrument (CREDI) Score (Long Form)
Biomarkers of micronutrient status, growth factors, systemic inflammation, environmental enteric dysfunction, metabolomics, choline, lipid panel (including HDL and LDL cholesterol) | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, at time of birth, and at 1 and 6 months post birth
  Measured using whole blood or serum samples among women and infants
Maternal blood pressure | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, at time of birth, and at 1 and 6 months post birth
  Diastolic and systolic blood pressure will be measured during pregnancy.

OTHER OUTCOMES:
Thalamus length | Between 20-26 weeks and 30-34 weeks gestational ages
  Thalamic measurements in cm, based on ultrasound
Thalamus width | Between 20-26 weeks and 30-34 weeks gestational ages
  Thalamic measurements in cm, based on ultrasound
Thalamus transverse | Between 20-26 weeks and 30-34 weeks gestational ages
  Thalamic measurements in cm, based on ultrasound
All-5 (indicator of eating all five food groups) | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, and at 1 and 6 months post birth
  Dietary Quality Questionnaire will be used to generate the All-5; range 0-5, where 5=1 and les than 5 = 0 (higher score, better outcome)
Animal Source Food Consumption | Between 9-<14 weeks, 20-26 weeks, and 30-34 weeks gestational ages, and at 1 and 6 months post birth
  Dietary Quality Questionnaire will be used to generate an indicator of animal source food consumption (milk, meat, eggs, fish), used here to generate a score (0-4), 4 is better.
Child motor development | 6 months of age
  Measured according to the Caregiver Reported Early Childhood Development Instrument (CREDI) Score, domain-specific motor development
Child cognitive development | 6 months of age
  Measured according to the Caregiver Reported Early Childhood Development Instrument (CREDI) Score, domain-specific cognitive development
Child social-emotional development | 6 months of age
  Measured according to the Caregiver Reported Early Childhood Development Instrument (CREDI) Score, domain-specific social-emotional development
Child language development | 6 months of age
  Measured according to the Caregiver Reported Early Childhood Development Instrument (CREDI) Score, domain-specific language development

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McKune, PhD, MPH, Principal Investigator — University of Florida
Locations (1):
- Ndama Health Center, Nyagatare, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Long-term preservation of the data Data will be de-identified and stored for future use after the completion of the study. The de-identified data set will not include any information that could lead to the identification of study participants, following the guidelines established by the HIPAA. Identifiable data will be destroyed after completion of the study. Long-term preservation of the de-identified data will ensure accessibility beyond the project's life.
  After the completion of the project, the de-identified data will be deposited into the Data Repository of the University of Florida and the USAID data repository, where it can be publicly accessed. Dataset in USAID repository will be findable and identifiable through a study digital object identifier (DOI).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 24 months after completion of the project
Access Criteria: the de-identified data will be deposited into the Data Repository of the University of Florida and the USAID data repository, where it can be publicly accessed. Dataset in USAID repository will be findable and identifiable through a study digital object identifier (DOI).

REFERENCES:
- [Background] Adu-Afarwuah S, Lartey A, Okronipa H, Ashorn P, Zeilani M, Peerson JM, Arimond M, Vosti S, Dewey KG. Lipid-based nutrient supplement increases the birth size of infants of primiparous women in Ghana. Am J Clin Nutr. 2015 Apr;101(4):835-46. doi: 10.3945/ajcn.114.091546. Epub 2015 Feb 11. PMID 25833980
- [Background] Adesogan, A. T., Havelaar, A. H., McKune, S. L., Eilittä, M., & Dahl, G. E. (2020). Animal source foods: Sustainability problem or malnutrition and sustainability solution? Perspective matters. Global Food Security, 25, 100325. https://doi.org/10.1016/j.gfs.2019.100325
- [Background] Christian P, Smith ER, Lee SE, Vargas AJ, Bremer AA, Raiten DJ. The need to study human milk as a biological system. Am J Clin Nutr. 2021 May 8;113(5):1063-1072. doi: 10.1093/ajcn/nqab075. PMID 33831952
- [Background] Cusick SE, Georgieff MK. The Role of Nutrition in Brain Development: The Golden Opportunity of the "First 1000 Days". J Pediatr. 2016 Aug;175:16-21. doi: 10.1016/j.jpeds.2016.05.013. Epub 2016 Jun 3. No abstract available. PMID 27266965
- [Background] Darapheak C, Takano T, Kizuki M, Nakamura K, Seino K. Consumption of animal source foods and dietary diversity reduce stunting in children in Cambodia. Int Arch Med. 2013 Jul 17;6:29. doi: 10.1186/1755-7682-6-29. eCollection 2013. PMID 23866682
- [Background] de Onis M, Branca F. Childhood stunting: a global perspective. Matern Child Nutr. 2016 May;12 Suppl 1(Suppl 1):12-26. doi: 10.1111/mcn.12231. PMID 27187907
- [Background] de Onis M, Onyango AW, Borghi E, Garza C, Yang H; WHO Multicentre Growth Reference Study Group. Comparison of the World Health Organization (WHO) Child Growth Standards and the National Center for Health Statistics/WHO international growth reference: implications for child health programmes. Public Health Nutr. 2006 Oct;9(7):942-7. doi: 10.1017/phn20062005. PMID 17010261
- [Background] Dhaded SM, Hambidge KM, Ali SA, Somannavar M, Saleem S, Pasha O, Khan U, Herekar V, Vernekar S, Kumar S Y, Westcott JE, Thorsten VR, Sridhar A, Das A, McClure E, Derman RJ, Goldenberg RL, Koso-Thomas M, Goudar SS, Krebs NF. Preconception nutrition intervention improved birth length and reduced stunting and wasting in newborns in South Asia: The Women First Randomized Controlled Trial. PLoS One. 2020 Jan 29;15(1):e0218960. doi: 10.1371/journal.pone.0218960. eCollection 2020. PMID 31995570
- [Background] Eaton JC, Rothpletz-Puglia P, Dreker MR, Iannotti L, Lutter C, Kaganda J, Rayco-Solon P. Effectiveness of provision of animal-source foods for supporting optimal growth and development in children 6 to 59 months of age. Cochrane Database Syst Rev. 2019 Feb 19;2(2):CD012818. doi: 10.1002/14651858.CD012818.pub2. PMID 30779870
- [Background] Ejigu H, Tafese Z. Stunting at birth: linear growth failure at an early age among newborns in Hawassa city public health hospitals, Sidama region, Ethiopia: a facility-based cross-sectional study. J Nutr Sci. 2023 May 30;12:e63. doi: 10.1017/jns.2023.46. eCollection 2023. PMID 37313345
- [Background] FAO (2001). Food and Report Technical Series Food and Energy Requirements. Retrieved from: https://www.fao.org/3/Y5686E/y5686e00.htm#Contentshttps://www.fao.org/3/Y5686E/y5686e00.ht m#Contents
- [Background] Fernandez ML. Eggs and health benefits. Can J Cardiol. 2011 Mar-Apr;27(2):264.e1; author reply 264.e7-8. doi: 10.1016/j.cjca.2010.12.014. No abstract available. PMID 21459286
- [Background] Giashuddin MS, Kabir M, Rahman A, Hannan MA. Exclusive breastfeeding and nutritional status in Bangladesh. Indian J Pediatr. 2003 Jun;70(6):471-5. doi: 10.1007/BF02723136. PMID 12921314
- [Background] Hahn, J., Dehghan, M., Drouin-Chartier, J. P., Mentz, R. J., Jneid, H., Virani, S. S., ... & Krittanawong, C. (2021). Egg consumption and risk of cardiovascular disease: A critical review. Current Emergency and Hospital Medicine Reports, 9, 25-37. https://doi.org/10.1007/s40138-021-00225-w
- [Background] Hambidge KM, Westcott JE, Garces A, Figueroa L, Goudar SS, Dhaded SM, Pasha O, Ali SA, Tshefu A, Lokangaka A, Derman RJ, Goldenberg RL, Bose CL, Bauserman M, Koso-Thomas M, Thorsten VR, Sridhar A, Stolka K, Das A, McClure EM, Krebs NF; Women First Preconception Trial Study Group. A multicountry randomized controlled trial of comprehensive maternal nutrition supplementation initiated before conception: the Women First trial. Am J Clin Nutr. 2019 Feb 1;109(2):457-469. doi: 10.1093/ajcn/nqy228. PMID 30721941
- [Background] Hendrixson DT, Smith K, Lasowski P, Callaghan-Gillespie M, Weber J, Papathakis P, Iversen PO, Koroma AS, Manary MJ. A novel intervention combining supplementary food and infection control measures to improve birth outcomes in undernourished pregnant women in Sierra Leone: A randomized, controlled clinical effectiveness trial. PLoS Med. 2021 Sep 28;18(9):e1003618. doi: 10.1371/journal.pmed.1003618. eCollection 2021 Sep. PMID 34582451
- [Background] Iannotti LL, Lutter CK, Stewart CP, Gallegos Riofrio CA, Malo C, Reinhart G, Palacios A, Karp C, Chapnick M, Cox K, Waters WF. Eggs in Early Complementary Feeding and Child Growth: A Randomized Controlled Trial. Pediatrics. 2017 Jul;140(1):e20163459. doi: 10.1542/peds.2016-3459. Epub 2017 Jun 7. PMID 28588101
- [Background] Imdad A, Bhutta ZA. Maternal nutrition and birth outcomes: effect of balanced protein-energy supplementation. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:178-90. doi: 10.1111/j.1365-3016.2012.01308.x. PMID 22742610
- [Background] Martorell R. Improved nutrition in the first 1000 days and adult human capital and health. Am J Hum Biol. 2017 Mar;29(2):10.1002/ajhb.22952. doi: 10.1002/ajhb.22952. Epub 2017 Jan 24. PMID 28117514
- [Background] McKune, S. L., Mechlowitz, K., & Miller, L. C. (2022). Dietary animal source food across the lifespan in LMIC. Global Food Security, 35, 100656. https://doi.org/10.1016/j.gfs.2022.100656
- [Background] McKune SL, Stark H, Sapp AC, Yang Y, Slanzi CM, Moore EV, Omer A, Wereme N'Diaye A. Behavior Change, Egg Consumption, and Child Nutrition: A Cluster Randomized Controlled Trial. Pediatrics. 2020 Dec;146(6):e2020007930. doi: 10.1542/peds.2020-007930. PMID 33239474
- [Background] MoH, Republic of Rwanda. (2019). Health sector performance report. https://www.moh.gov.rw/fileadmin/user_upload/Moh/Publications/Reports/Health_Sector_Annual_P erformance_Report_2020-2021.pdf
- [Background] Murphy SP, Allen LH. Nutritional importance of animal source foods. J Nutr. 2003 Nov;133(11 Suppl 2):3932S-3935S. doi: 10.1093/jn/133.11.3932S. PMID 14672292
- [Background] Myers M, Ruxton CHS. Eggs: Healthy or Risky? A Review of Evidence from High Quality Studies on Hen's Eggs. Nutrients. 2023 Jun 7;15(12):2657. doi: 10.3390/nu15122657. PMID 37375561
- [Background] Namirembe G, Ghosh S, Ausman LM, Shrestha R, Zaharia S, Bashaasha B, Kabunga N, Agaba E, Mezzano J, Webb P. Child stunting starts in utero: Growth trajectories and determinants in Ugandan infants. Matern Child Nutr. 2022 Jul;18(3):e13359. doi: 10.1111/mcn.13359. Epub 2022 Apr 29. PMID 35488408
- [Background] Omer, A., Mulualem, D., Classen, H., Vatanparast, H., & Whiting, S. J. (2018). A community poultry intervention to promote egg and eggshell powder consumption by young children in Halaba Special Woreda, SNNPR, Ethiopia. J Agric Sci, 10(5), 1. https://doi.org/10.5539/jas.v10n5p1
- [Background] Picciano MF. Pregnancy and lactation: physiological adjustments, nutritional requirements and the role of dietary supplements. J Nutr. 2003 Jun;133(6):1997S-2002S. doi: 10.1093/jn/133.6.1997S. PMID 12771353
- [Background] Republic of Rwanda MOH, Rwanda Biomedical Centre, National Child Development Agency. Report of Maternal and Child Health Week Campaign, May 16-20, 2022. Kigali, Rwanda: MOH. 2022:25.
- [Background] Santosa A, Novanda Arif E, Abdul Ghoni D. Effect of maternal and child factors on stunting: partial least squares structural equation modeling. Clin Exp Pediatr. 2022 Feb;65(2):90-97. doi: 10.3345/cep.2021.00094. Epub 2021 May 4. PMID 33957035
- [Background] Schwarzenberg SJ, Georgieff MK; COMMITTEE ON NUTRITION. Advocacy for Improving Nutrition in the First 1000 Days to Support Childhood Development and Adult Health. Pediatrics. 2018 Feb;141(2):e20173716. doi: 10.1542/peds.2017-3716. Epub 2018 Jan 22. PMID 29358479
- [Background] Stevens B, Buettner P, Watt K, Clough A, Brimblecombe J, Judd J. The effect of balanced protein energy supplementation in undernourished pregnant women and child physical growth in low- and middle-income countries: a systematic review and meta-analysis. Matern Child Nutr. 2015 Oct;11(4):415-32. doi: 10.1111/mcn.12183. Epub 2015 Apr 7. PMID 25857334
- [Background] Stewart CP, Caswell B, Iannotti L, Lutter C, Arnold CD, Chipatala R, Prado EL, Maleta K. The effect of eggs on early child growth in rural Malawi: the Mazira Project randomized controlled trial. Am J Clin Nutr. 2019 Oct 1;110(4):1026-1033. doi: 10.1093/ajcn/nqz163. PMID 31386106
- [Background] Wang K, Xiang Q, Hu L, Wang L, Zhang Y. Frequency of Egg Intake Associated with Mortality in Chinese Adults: An 8-Year Nationwide Cohort Study. Int J Environ Res Public Health. 2022 Nov 10;19(22):14777. doi: 10.3390/ijerph192214777. PMID 36429496
- [Background] Zhang X, Lv M, Luo X, Estill J, Wang L, Ren M, Liu Y, Feng Z, Wang J, Wang X, Chen Y. Egg consumption and health outcomes: a global evidence mapping based on an overview of systematic reviews. Ann Transl Med. 2020 Nov;8(21):1343. doi: 10.21037/atm-20-4243. PMID 33313088
- [Derived] Tiwari C, Acosta D, Matsiko E, Kampire A, Nsabimana A, Stark H, Laborde JEA, Yang Y, Reider K, Nsereko E, Kirby M, McKune S. Deux Oeufs: cracking the potential of eggs to improve child growth and development - a randomized controlled trial (RCT) study protocol. Trials. 2025 Dec 23;26(1):578. doi: 10.1186/s13063-025-09237-3. PMID 41437064